CLINICAL TRIAL: NCT04703179
Title: Rare and Undiagnosed Disease Research Biorepository
Acronym: PRaUD
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Filippo Pinto e Vairo, Principal Investigator, Mayo Clinic
Other Study IDs: 19-003389
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Undiagnosed Disease; Rare Diseases
MeSH Terms: conditions — Undiagnosed Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Research blood collections kits will attempt to be collected on all active study participants. Other samples including urine, stool, tissue, fibroblasts, CSF, RNA, DNA and saliva may also be collected under the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Genetic test evaluation — Patients with rare and undiagnosed disease and their family members may be evaluated on a case by case basis. The research study may perform multi-omics testing to provide a diagnosis or to provide biomarker discovery.

SUMMARY:
This research study is being done to find markers and identify causes of rare and undiagnosed diseases by analyzing patient's DNA (i.e., genetic material), RNA, plasma, urine, tissues, or other samples that could be informative of symptoms. Researchers are creating a biobank (library) of samples and information to learn more about treating rare and undiagnosed diseases.

ELIGIBILITY:
Inclusion Criteria:

* Has Mayo Clinic or other medical health system ID, or another unique identifier
* Able to provide informed consent

Must meet one of the following:

* Individual must have evidence of a rare disease or a suspected genetic disorder as determined by a provider or genetic counselor
* Biological family member of an enrolled individual

Exclusion Criteria:

* Individuals who have situations that would limit compliance with the study requirements
* Institutionalized (i.e. Federal Medical Prison)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with any rare and undiagnosed disease. Both affected and unaffected family members may also be invited for participation as part of the genetic evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Enrollment of Study Participants | 5 years
  5,000 participants to be accrued

SECONDARY OUTCOMES:
Body-of-Knowledge | 5 years
  To prospectively follow the cohort of Rare and Undiagnosed Disease Biorepository participants to ascertain new health outcomes via medical records and patient contact, update risk factor data, and collect additional biologic specimens.
Discovery of Disease Mechanisms and Therapeutic Approaches | 5 years
  To facilitate research projects using the Rare and Undiagnosed Disease Biobank to identify underlying disease mechanisms and potential therapeutic approaches.
Diagnostic Yield | 5 years
  To change the rate of diagnosis and level of care for patients with rare and undiagnosed diseases through collaborations with clinical investigators and researchers at Mayo Clinic and globally.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pinto e Vairo, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials